CLINICAL TRIAL: NCT05785546
Title: Wheelchair Seating Users With Neuromuscular Diseases: Elaboration of a Pronostic Score of Changes on the Seating System of the Wheelchair
Brief Title: Elaboration of a Pronostic Score of Changes on Wheelchair's Seating System
Acronym: BPIP-Score MNM
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP210996; 2023-A00831-44 (Registry Identifier: IDRCB)
Record Dates: First submitted 2023-03-15; First posted 2023-03-27 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Neuromuscular Diseases
Keywords: Neuromuscular Diseases
MeSH Terms: conditions — Neuromuscular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- development cohort: Neuromuscular diseases
  Interventions: Other: usual care
- validation cohort: Neuromuscular diseases
  Interventions: Other: usual care

INTERVENTIONS:
Other: usual care — For each cohort, the patient is seen at least twice, during annual visits in multidisciplinary consultation.

SUMMARY:
Development and validation study of a prognostic score - study of prognostic performance by a prospective longitudinal multicenter cohort spread over 8 centers: 4 for the development cohort and 4 for the validation cohort).

DETAILED DESCRIPTION:
Progressive muscle weakness in neuromuscular diseases leads to motor disabilities leading to permanentfull-time wheelchair use. This is the case for infantile spinal muscular atrophy type II (SMA II), where people are dependent on a permanent sitting position from early childhood, at 2 years of age, or for Duchenne muscular dystrophy, when they lose their ability to walk around 10 years without corticosteroid therapy or around 13 years with treatment. These wheelchair users, weakened by the disease, are subject to musculotendinous retractions, osteo-articular stiffness, spinal deformities and pain. In addition, they use the wheelchair on a daily basis, on average 12 hours a day, whose permanent sitting position also conditions the performance of achieving life habits.

The analysis of the static and dynamic seated postural installation in the wheelchair makes it possible to avoid harmful consequences on the health and quality of life of users on a daily basis. When performed early enough, regularly and optimally, it also contributes to the prevention of complications.

In France, these assessments are carried out by occupational therapists, accompanied by doctors of Physical Medicine and Rehabilitation.

The weakness of the literature in this area and the absence of recommendations do not allow the user or any health professional to identify the need and the level of urgency to benefit from a dedicated consultation.

Faced with this observation, the development of a prognostic score for a change in positioning in the wheelchair, based on a prospective multicenter cohort and its validation on an external prospective cohort, will allow any healthcare professional to guide the user to a necessary positioning consultation. The hypothesis is that this score has discriminating qualities and that it is calibrated to predict a change in the seat of the RF and therefore the need to reassess the seated postural installation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over the age of 18
* Daily wheelchair user (more than 4 hours per day)
* Having a neuromuscular disease such as Duchenne Muscular Dystrophy or Infantile Spinal Muscular Atrophy type II
* Accompanied by an identified medical equipment provider, able to respond to the recommendations of the clinical team
* Patient informed and having signed consent.

Exclusion Criteria:

* Person who already has a seat change or FR prescription at the time of inclusion
* Having undergone surgery less than 1 year ago or a fracture
* Pregnant or breastfeeding women
* Patient under guardianship or curatorship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Having a neuromuscular disease such as Duchenne Muscular Dystrophy or Infantile Spinal Muscular Atrophy type II.
Sampling Method: Non-Probability Sample
Enrollment: 368 (Estimated)
Dates: Start 2025-02-19 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Change in the seating system of the user's wheelchair | through study completion, to 12 months
  Any change in the seating system of the user's wheelchair within 12 months will be noted.
  A change in the seating system is defined by the occurrence of at least one of these situations:
  * one or more seat/back adjustments: depth, width, height
  * addition/removal of postural elements
  * replacement of the cushion, or backrest or headrest
  * Use of electric functions of the wheelchair or on-board standing
  * modification of control device of the WC.

SECONDARY OUTCOMES:
Seated Postural Control Measure (SPCM) | at baseline and 12 months
  Seated Postural Control Measure (SPCM) is an instrument for the clinical assessment of seated postural control in adult clients using a locomotion aid. It therefore allows the evaluation of the two variables in inherent to postural control seated, i.e. the alignment of body segments and the influence between movement and posture. It also helps to assess changes of seated postural control due to the evolution over time or to an intervention of a adaptation of the sitting posture.
Pain Visual Analogue Scale | at baseline and 12 months
  To assess pain, the investigators will use a Visual Analog Scale (0-10).
Pressure ulcer topography (stage and location ) | at baseline and 12 months
  International NPUAP/EPUAP Pressure injury classification system
Comfort perception scale (Visual Analogue Scale) | at baseline and 12 months
  Visual Analog Scale (0-10) will be used to assess comfort of patients.
Postural stability perception scale (in antero-posterior and lateral stability) | at baseline and 12 months
  self-questionnaire will be used.
adverse event | through study completion, an average of 12 month
  Semi-structured interview following the identification of an adverse event in wheelchair by the user, within 12 months after inclusion.
  explain or understand the identification or not of an adverse event in wheelchair and its escalation to the clinical team, by the user.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Pouplin, PhD, Principal Investigator — New technology Platform department, Raymond Poincaré Hospital, APHP
Locations (1):
- New technology Platform department, Raymond Poincaré Hospital, APHP, Garches, France